CLINICAL TRIAL: NCT03149055
Title: A Single Center, Open-label Trial of Isavuconazole Prophylaxis Against Invasive Fungal Infection in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplant (HCT)
Brief Title: Fungal Prophylaxis With Isavuconazole for Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplant (HCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-112
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Results first posted 2020-08-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2021-11

CONDITIONS: Hematologic Malignancy; Myeloproliferative Disorder
MeSH Terms: conditions — Hematologic Neoplasms; Myeloproliferative Disorders | interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isavuconazole prophylaxis (Experimental): Intravenous or oral: Isavuconazonium sulfate 372 mg Q 8hour for 6 doses as loading dose, followed by 372 mg Q day as maintenance dose. The minimum duration of prophylaxis with isavuconazole will be through D +60. Beyond day +60 discontinuation is at the discretion of the treating physician.
  Interventions: Drug: Isavuconazole

INTERVENTIONS:
Drug: Isavuconazole — Intravenous or oral: Isavuconazonium sulfate 372 mg Q 8hour for 6 doses as loading dose, followed by 372 mg Q day as maintenance dose.
  Other Names: Isavuconazonium sulfate

SUMMARY:
The purpose of this study is to study the effects of isavuconazole in preventing fungal infections in patients who have had a hematopoietic stem cell transplant (HCT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of greater than or equal to 18 years of age of either sex and of any race.
* Have received first peripheral blood, marrow or cord blood transplant from a family or unrelated donor for hematologic malignancy or myeloproliferative disorder.

Exclusion Criteria:

* Proven or probable aspergillosis or other mold infection or deep mycoses including hepatosplenic candidiasis less than 60 days from first dose of ISA.
* History of allergy or intolerance to ISA.
* Clinically significant elevation of liver function tests prior to the first day of dosing (FDD) that at the discretion of the treating physician would preclude the administration of an azole antifungal.
* Familial short QT syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2021-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isavuconazole Prophylaxis
Started | 99
Completed | 95
Not Completed | 4
Not completed — Not treated | 4

BASELINE CHARACTERISTICS:
Arm/Group | Isavuconazole Prophylaxis
Number analyzed (Participants) | 95
Age, Continuous [Median (Full Range); unit: years] | 57 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 81
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95
Underlying Disease [Count of Participants; unit: Participants]
  Leukemia | 51
  Myelodysplastic syndrome | 15
  Lymphoma | 16
  Other hematologic malignancy | 13
Graft Manipulation [Count of Participants; unit: Participants]
  Ex vivo T-cell depletion (CD4+ selected) | 31
  No graft manipulation | 64
Donor Type [Count of Participants; unit: Participants]
  Matched related | 19
  Matched unrelated | 36
  Mismatched related/unrelated | 26
  Haploidentical | 14
Hematopoietic cell transplant (HCT) Source [Count of Participants; unit: Participants]
  Peripheral blood (PBSC) | 64
  Bone marrow | 17
  Cord blood | 14
Conditioning Regimen Intensity [Count of Participants; unit: Participants]
  Myeloablative | 53
  Non-myeloablative | 13
  Reduced intensity | 29
Graft versus Host Disease (GvHD) Prophylaxis [Count of Participants; unit: Participants] — *7 patients also received sirolimus in addition to tacrolimus and methotrexate
  **11 patients received tocilizumab in addition to Cyclosporine + MMF
  Cyclophosphamide + Mycophenolate + Tacrolimus or Sirolimus***
  ***Cyclophosphamide was administered post HCT. Tacrolimus (19 patients); Sirolimus (3 patients)
  Participants
    Tacrolimus + Methotrexate* | 26
    Cyclosporine + Mycophenolate Mofetil** | 16
    Tacrolimus + Mycophenolate Mofetil | 2
    Cyclophosphamide+Mycophenolate+Tacrolimus or Si*** | 22
    Ex vivo T-cell depletion | 29

OUTCOME MEASURES:

1. Primary Outcome: Clinical Failure of Isavuconazole Prophylaxis by Week + 14 Post Hematopoietic Stem Cell Transplant (HCT)
Description: Clinical failure is measured by:
  1. Systemic antifungal therapy for > 14 consecutive days for suspected fungal infection up to week 14.
  2. Breakthrough proven or probable fungal infection during the prophylaxis phase.*
  3. Toxicity leading to permanent discontinuation of prophylaxis
  4. Adverse event requiring discontinuation.
     * The prophylaxis phase was defined as the period from the first dose of isavuconazole through 7 days after discontinuation of isavuconazole.
Time Frame: 14 weeks post HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Isavuconazole Prophylaxis
Number analyzed (Participants) | 95
Participants
  Completed Treatment | 81
  Did not complete treatment, breakthrough IFI | 3
  Did not complete treatment, discont d/t toxicity | 7
  Did not complete treatment, other reasons | 4

2. Primary Outcome: Clinical Failure of Isavuconazole Prophylaxis by Week + 26 Post Hematopoietic Stem Cell Transplant (HCT)
Description: as for outcome 1
Time Frame: 26 weeks post HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Isavuconazole Prophylaxis
Number analyzed (Participants) | 95
Participants
  Completed Study | 89
  Did Not Complete Study d/t Death | 6

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: AE's leading to Isavuconazole discontinuation were collected
Arm/Group | Isavuconazole Prophylaxis
All-Cause Mortality (participants affected / at risk) | 6/95
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 7/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Isavuconazole Prophylaxis (N=95)
Rash (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Transaminitis (Hepatobiliary disorders) | 2
Hyperbilirubinemia (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT03149055/Prot_SAP_000.pdf